CLINICAL TRIAL: NCT02646410
Title: Optimal Delivery of Seasonal Malaria Chemoprevention and Its Effects on the Acquisition of Malaria Immunity
Brief Title: Optimization of Seasonal Malaria Chemoprevention (SMC) Delivery
Acronym: SMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bamako (Other)
Responsible Party: Principal Investigator, Alassane Dicko, Professor, University of Bamako
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2014-61
Record Dates: First submitted 2015-12-29; First posted 2016-01-05 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Malaria; Anemia
Keywords: malaria; seasonal malaria chemoprevention; immunity; resistance; sulfadoxine-pyrimethamine; amodiaquine; delivery method
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- FPD+NDOT (Other): Fixed-point delivery (FPD) combined with non directly observed treatment (NDOT)
  Interventions: Other: FPD+NDOT
- FPD+DOT (Other): Fixed-point delivery (FPD) combined with directly observed treatment (DOT)
  Interventions: Other: FPD+DOT
- DDD+NDOT (Other): door-to-door delivery (DDD) combined with non directly observed treatment (NDOT)
  Interventions: Other: DDD+NDOT
- DDD+DOT (Other): door-to-door delivery (DDD) combined with directly observed treatment (NDOT)
  Interventions: Other: DDD+DOT

INTERVENTIONS:
Other: FPD+NDOT
  Other Names: fixed-point delivery + non directly observed treatment
  Arms: FPD+NDOT
Other: FPD+DOT
  Other Names: fixed-point delivery + directly observed treatment
  Arms: FPD+DOT
Other: DDD+NDOT — Door to door delivery + non directly observed treatment
  Arms: DDD+NDOT
Other: DDD+DOT — Door to door delivery + directly observed treatment
  Arms: DDD+DOT

SUMMARY:
Based in part on the pivotal studies conducted in Mali, SMC was approved by WHO as a policy for malaria control in countries with seasonal malaria transmission such as Mali in March 2012. The goals are to identify the most effective method to deliver SMC, and to obtain more information on the long term impact of SMC on malaria immunity. Our specific aims are 1) to determine the optimal mode (fixed-point (FPD) vs door-to-door delivery (DDD); directly observed treatment (DOT) vs non-DOT (NDOT)) and frequency (3 vs 4 doses per season) of SMC delivery; 2) to compare quantitative measures of immunity in children who do and do not receive SMC. A cluster-randomized design will be sued. The target population will be children aged 3-59 months old in Ouelessebougou district, Mali. In Year 1, villages in four sub-districts will be randomized into four groups (FPD+DOT; FPD+NDOT; DDD+DOT; DDD+NDOT). The optimal mode of delivery will be selected based on the SMC coverage during the first year, and will then be implemented in villages of two additional sub-districts. Villages in these two newly selected sub-districts will be randomized in two groups. Children in the first group will received three rounds of SMC and those in the second group will receive four rounds of SMC to determine the optimal frequency of SMC based on the incidence rate of clinical malaria as measured by passive surveillance. In Year 3, children in the selected sub-districts will received SMC by the optimal delivery system determined in Years 1 -2. A survey will be conducted collect data on mortality and hospital admission and compare these outcomes in areas where SMC was implemented and areas where SMC was not implemented.

DETAILED DESCRIPTION:
Based in part on the pivotal studies conducted in Mali, SMC was approved by WHO as a policy for malaria control in countries with seasonal malaria transmission such as Mali in March 2012. The strategy is a highly cost-effective approach to reduce childhood mortality in these areas. Despite the huge benefit of the SMC on malaria infection and disease, the optimal approach to deliver SMC remains to be determined and there is no data on the long term effect of this strategy on the development of immunity to malaria. While fixed-point delivery (FPD) combined with non directly observed treatment (NDOT) by community health workers is attractive for the SMC implementation, it is need to be evaluated and compared to other mode of delivery. The objectives are to identify the most effective method to deliver SMC, and to obtain information on the long term impact of SMC on malaria immunity. Specifically, i) to determine the optimal mode (fixed-point (FPD) vs door-to-door delivery (DDD); directly observed treatment (DOT) vs. non-DOT (NDOT)) and frequency (3 vs. 4 doses per season) of SMC delivery; ii) to compare quantitative measures of immunity in children who do and do not receive SMC over a three year period.

The design is a cluster-randomized trial over three years. The target population is children aged 3-59 months old living in Ouelessebougou district, Mali. In Year 1, villages in four sub-districts will be randomized into four groups (FPD+DOT; FPD+NDOT; DDD+DOT; DDD+NDOT). The optimal mode of delivery will be selected based on the SMC coverage during the first year, and will then be implemented in villages of two additional sub-districts. Villages in these two newly selected sub-districts will be randomized in two groups. Children in the first group will received three rounds of SMC and those in the second group will receive four rounds of SMC to determine the optimal frequency of SMC based on the incidence rate of clinical malaria as measured by passive surveillance. Children in the four sub-districts selected in Year 1 will continue to receive three rounds of SMC in Year 2 using the optimal mode of delivery. In Year 3, children in the randomly selected sub-districts will received SMC by the optimal delivery system determined in Years 1 -2. Immune responses will be measured and compared between the children receiving SMC to a cohort of children not receiving SMC, to assess the impact of SMC on key antimalarial antibody responses over the three year period using cross-sectional surveys at the beginning and the end of the transmission season.

In Year 3, 4 and 5 surveys will be conducted to collect data on mortality and hospital admissions and compare these outcomes in areas where SMC was implemented and areas where SMC was not implemented.

ELIGIBILITY:
Inclusion Criteria:

Age >= 3 months & < 60 months

Exclusion Criteria:

* severe, chronic illness
* known allergy to one of the study drugs (SP or AQ)
* known HIV positive subjects using Cotrimoxazole.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10000 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Coverage of SMC | 1-5 weeks after last round of SMC in Year1
  SMC coverage will be defined as proportion of the children who have received the three treatments doses at each of the three rounds of SMC.
Incidence of clinical malaria in Year 2 | up to 4 weeks after the last round of SMC
  Clinical malaria defined as signs and symptoms suggestive of malaria with positive RDT and/or positive blood smear.
Mortality rate | 1, 2, 3, 4 years of the intervention
  death
Hospital admission | 1, 2, 3, 4 years of the intervention
  Hospitalization

SECONDARY OUTCOMES:
malaria parasitemia | one week before the first round of SMC and 4-6 weeks after the last round of SMC
  Parasite prevalence defined as the proportion of children with a positive malaria blood smear and parasite density
moderate anemia | one week before the first round of SMC and 4-6 weeks after the last round of SMC
  Prevalence of moderate anemia defined as hemoglobin concentration < 8 g/dL measured by hemoglobin analyzer
immune response to malaria parasite | one week before the first round of SMC and 4-6 weeks after the last round of SMC
  Cellular and humoral antimalarial immune responses to malaria parasites
molecular markers of resistance to SP + AQ | one week before the first round of SMC and 4-6 weeks after the last round of SMC
  Frequency of mutations at codons 51, 59, and 108 of the dhfr gene, 437 and 540 of the dhps gene, codon 76 in the P. falciparum chloroquine transporter gene (pfcrt), and codon 86 of the P. falciparum multidrug resistance gene one (pfmdr1).
nutritional status | one week before the first round of SMC and 4-6 weeks after the last round of SMC
  Prevalence of wasting stunting and underweight as defined by WHO Global database on Child Growth and Malnutrition
Clinical malaria in Year 1 | up to 4 weeks after the last round of SMC
  Clinical malaria defined as signs and symptoms suggestive of malaria with positive RDT and/or positive blood smear.

CONTACTS AND LOCATIONS:
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Derived] Issiaka D, Barry A, Traore T, Diarra B, Cook D, Keita M, Sagara I, Duffy P, Fried M, Dicko A. Impact of seasonal malaria chemoprevention on hospital admissions and mortality in children under 5 years of age in Ouelessebougou, Mali. Malar J. 2020 Mar 3;19(1):103. doi: 10.1186/s12936-020-03175-y. PMID 32126989
- [Derived] Barry A, Issiaka D, Traore T, Mahamar A, Diarra B, Sagara I, Kone D, Doumbo OK, Duffy P, Fried M, Dicko A. Optimal mode for delivery of seasonal malaria chemoprevention in Ouelessebougou, Mali: A cluster randomized trial. PLoS One. 2018 Mar 5;13(3):e0193296. doi: 10.1371/journal.pone.0193296. eCollection 2018. PMID 29505578